CLINICAL TRIAL: NCT05483257
Title: Molecular Subtyping Based on Specific HLA-I Genotypes for Prognosis Evaluation in Resected Pancreatic Adenocarcinoma: A Retrospective Observational Cohort Study
Brief Title: Molecular Subtyping for Prognosis Evaluation in Resected Pancreatic Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: BAIYONG SHEN (Other)
Collaborators: GeneCast Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, BAIYONG SHEN, Professor, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Other Study IDs: M-Cli200633-PC
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Pancreatic Cancer Resectable
Keywords: human leukocyte antigen class I; supertypes; recurrence
MeSH Terms: conditions — Recurrence | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Matched blood cells and tumor tissues
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Multigene panel for next-generation sequencing — HLA-I genotyping based on next-generation sequencing for prognosis evaluation

SUMMARY:
Pancreatic adenocarcinoma (PAAD) patients following surgeries are prone to relapse shortly, while it is not well understood by current biomarkers. Given the potential associations of human leukocyte antigen class I (HLA-I) genotype with oncogenic mutational profile and immunotherapy efficacy, we aimed to assess whether differential HLA-I genotype could predict the postoperative outcomes in resected PAAD patients.

ELIGIBILITY:
Inclusion Criteria:

* Radically resected pancreatic adenocarcinoma (stage I-III)
* Resected tumor tissues and matched blood cells available
* Signed informed consent

Exclusion Criteria:

* Pancreatic cancer except pancreatic adenocarcinoma
* Non-radical resection

Ages: 34 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Radically resected patients with pancreatic adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 2 years
  Comparison of DFS between patients with specific HLA-I genotypes or not

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wen C, Zhang L, Yang Y, Jin Y, Ren D, Zhang Z, Zou S, Li F, Sun H, Jin J, Lu X, Xie J, Cheng D, Xu Z, Chen H, Mao B, Zhang J, Wang J, Deng X, Peng C, Li H, Jiang C, Lin L, Zhang H, Chen H, Shen B, Zhan Q. Specific human leukocyte antigen class I genotypes predict prognosis in resected pancreatic adenocarcinoma: a retrospective cohort study. Int J Surg. 2023 Jul 1;109(7):1941-1952. doi: 10.1097/JS9.0000000000000264. PMID 37026827